CLINICAL TRIAL: NCT03628261
Title: Is EMG-based Serious Games Effective in Improving Gait in Children With Cerebral Palsy ? Interest of Electromyography Feedback (EMG)
Acronym: SERIOUS GAME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2017-63; 2018-A00831-54 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- physical therapy then serious games (Other): Children will receive four weeks of treatment with EMG-based serious games in addition to the conventional physiotherapy
  Interventions: Device: Serious Game; Other: physical therapy
- serious games then physical therapy (Other): Children will receive four weeks of treatment with EMG-based serious games in addition to the conventional physiotherapy
  Interventions: Device: Serious Game; Other: physical therapy

INTERVENTIONS:
Device: Serious Game — Surface EMG detection for the myoelectric control of the EMG-based serious games and for the EMG assessment during gait will be performed with a wireless system.This device is composed of seven modules (sensor units), each detecting and transmitting two bipolar EMGs at 2 kilo Hertz (kHz). During the evaluation protocol EMGs will be detected from peroneus longus, gastrocnemius medialis, soleus and tibialis anterior muscles of both limbs using pre-gelled electrodes.
Other: physical therapy — Children receive the regular rehabilitation for the treatment of ankle plantar flexor muscle overactivity and the paresis of ankle dorsal flexor muscle

SUMMARY:
Cerebral palsy (CP) is a major motor dysfunction manifesting early in childhood, with severe consequences to performance in daily functions. CP children are typically unable to voluntarily activate individual muscles, hindering motor coordination and therefore the ability to produce movements as smooth as those seen in control cohorts. Muscles spanning distal joints are more likely affected by CP, resulting in abnormal gait patterns.

While commercially available and customised games have been considered for CP rehabilitation in the last decade, they are mainly based on the analysis of movement kinematics and none seems to deal directly with the key source of motor impairment: the skeletal muscle. Surface electromyograms (EMGs), on the other hand, provide clinicians with the possibility of directly assessing and controlling the neural drive or command to muscles.

The benefits of surface EMG as a feedback tool for improving posture control and for stroke rehabilitation are well established.

The treatment with EMG-based "serious games" is expected to assist CP children in activating the ankle muscles in both paretic and healthy limbs at similar instants within the gait cycle. Given such EMG-oriented rehabilitation applies directly to the muscle, its effect on muscle and therefore gait function is likely to be greater than that achieved with conventional means. If this hypothesis is verified, it will be further expect to observe a smoother gait, that is smoother changes in gait kinematics and morphology of the paretic foot, in CP children treated with EMG-based serious game than otherwise.

Primary objective consists in verifying whether Surface electromyography (sEMG)-based games are effective in reducing the degree of muscular hyperactivity in the ankle plantar flexor and thus improve the ankle dorsi flexor function in children with cerebral palsy.

The study design is an open, prospective, monocentric, randomized and controlled trial. Participants will be randomly assigned to either the first group or to the second group.

For the first group, the design will be: "physical therapy + serious games" during the first month then "physical therapy" during the second month.

For second group, the the design will be: "physical therapy" during the first month then "physical therapy + serious games" during the second month.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 2 to 10 years,
* Hemiparetic child (left or right) by cerebral palsy, (scoring Level 1 or 2 on the Gross Motor Function Classification System),
* Initial contact during gait (just before the stance phase) with Equinovarus or Equinovalgus ,
* Child with cognitive functions compatible with the instructions of serious games,
* Children with parents (or legal guardians) authorizing participation in the study and a signed informed consent form,
* Children affiliated with medical insurance.

Exclusion Criteria:

* Children under 2 years old and over 10 years old,
* Children who have had orthopedic surgery and / or administration of botulinum toxin to the calf muscles within six months prior to study participation.

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-01-04 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
number of muscle was activated during gait | 12 months
  Onsets of muscle activation will be estimated using a semi-automated method, with activation instants being defined by when the rectified, raw EMG exceeds 20 millivolt (mV). The timing of muscle activity will be expressed as a percentage of gait cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Olivier ARNAUD, Director, Study Director — Assistance Publique des Hôpitaux de Marseille
Locations (1):
- Assistance Publique Hôpitaux de Marseille, Marseille, France

IPD SHARING:
Plan to Share IPD: No